CLINICAL TRIAL: NCT02146365
Title: A Prospective Study to Assess the Nasopharyngeal Carriage of Streptococcus Pneumoniae (SPn), Long Term Safety and Immune Persistence in Healthy Kenyan PCV-Primed Toddlers (12-15 Months of Age) Who Received a Whole Cell Pneumococcal Vaccine (PATH-wSP) Compared to Controls
Brief Title: Nasopharyngeal Carriage Study in Healthy Kenyan Toddlers
Status: Completed | Type: Observational
Sponsor: PATH (Other)
Responsible Party: Sponsor
Other Study IDs: VAC-011
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-01

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasal swab sample and blood draw
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- PATH-wSP 300 µg + Booster: Toddlers who enrolled in Cohort 1 of Study VAC-010 and received 300 µg PATH-wSP plus the two booster vaccines (Synflorix and Pentavac) followed by a 2nd injection of 300 µg PATH-wSP 8 weeks later.
- PATH-wSP 300 µg Only: Toddlers who enrolled in Cohort 1 of Study VAC-010 and received 300 µg PATH-wSP and 2 saline injections followed by a 2nd injection of 300 µg PATH-wSP 8 weeks later.
- PATH-wSP 600 µg + Booster: Toddlers who enrolled in Cohort 2 of Study VAC-010 and received 600 µg PATH-wSP plus the two booster vaccines (Synflorix and Pentavac) followed by a 2nd injection of 600 µg PATH-wSP 8 weeks later.
- PATH-wSP 600 µg Only: Toddlers who enrolled in Cohort 2 of Study VAC-010 and received 600 µg PATH-wSP and 2 saline injections followed by a 2nd injection of 600 µg PATH-wSP 8 weeks later.
- Booster Only (300 µg): Toddlers who enrolled in Cohort 1 of Study VAC-010 and received one saline injection and the two booster vaccines (Synflorix and Pentavac) followed by a 2nd saline injection 8 weeks later.
- Booster Only (600 µg): Toddlers who enrolled in Cohort 2 of Study VAC-010 and received one saline injection and the two booster vaccines (Synflorix and Pentavac) followed by a 2nd saline injection 8 weeks later.
- No Intervention (300 µg): Toddlers who enrolled during Cohort 1 who did not participate in Study VAC-010 and did not receive either PATH-wSP or either of the booster vaccines (Pentavac or Synflorix).
- No Intervention (600 µg): Toddlers who enrolled during Cohort 2 who did not participate in Study VAC-010 and did not receive either PATH-wSP or either of the booster vaccines (Pentavac or Synflorix).

SUMMARY:
This study evaluated the change in nasopharyngeal carriage (NPC) of Streptococcus pneumoniae (SPn), hypothesizing that it would be reduced post-vaccination with Streptococcus pneumoniae whole cell vaccine with aluminum hydroxide adjuvant (PATH-wSP) and that PATH-wSP would remain safe and well-tolerated over the course of the study.

DETAILED DESCRIPTION:
This study enrolled healthy Kenyan toddlers (12-15 months of age) who participated in the randomized control trial of VAC-010 (NCT02097472), as well as healthy toddlers aged 12 to 15 months who had not participated in the VAC-010 Study. All participants must have received a primary dose of pneumococcal conjugate vaccine (PCV) per local practice prior to enrollment in either VAC-010 or VAC-011. No treatments were administered during this study.

The study consisted of the following four groups:

Participants who were randomized in study VAC-010 (2:2:1 ratio), defined according to the treatment received in VAC-010:

* 1. PATH-wSP + Booster
* 2. PATH-wSP Only
* 3. Booster Only

Participants who did not participate in VAC-010:

* 4. No Intervention

Each group consisted of 2 cohorts of participants, Cohort 1 (300 µg PATH-wSP) and Cohort 2 (600 µg PATH-wSP). Enrollment into Cohorts 1 and 2 occurred sequentially; participants in groups 3 and 4 who did not receive PATH-wSP were also enrolled over time and allocated into one of the two cohorts (300 and 600 µg) in order to control for potential seasonal variation in the NPC of S. pneumoniae.

Each participant completed a total of 5 scheduled visits. For toddlers enrolled simultaneously in VAC-010, visits corresponded to enrollment (Baseline) and 4, 8, 12, and 24 weeks post final vaccination in VAC-010. For toddlers in the No Intervention group, the first visit corresponded to Baseline and the second to fifth visits corresponded to 12, 16, 20, and 32 weeks later. Nasopharyngeal swabs were taken at each visit following World Health Organization (WHO) guidelines for analysis of nasopharyngeal burden.

Treatments received during VAC-010 included:

* PATH-wSP: Streptococcus pneumoniae whole cell vaccine with aluminum hydroxide adjuvant
* Synflorix™ booster vaccine: pneumococcal polysaccharide conjugate vaccine (adsorbed)
* Pentavac booster vaccine: diphtheria, tetanus, pertussis (Whole Cell), hepatitis B (recombinant deoxyribonucleic acid [rDNA]) and Haemophilus influenzae type b conjugate vaccine (adsorbed).
* Saline control

ELIGIBILITY:
Inclusion Criteria:

- For Toddlers Enrolled in VAC-010 (NCT02097472):

* Randomization in VAC-010.
* Subject's parent must provide voluntary written informed consent for subject to participate in the study, is fully capable of comprehending and complying with study requirements and procedures, able and willing to return for all scheduled follow-up visits, and has expressed availability for the required study period, with access to a consistent means of telephone contact. An illiterate parent will require an impartial witness to be present during consenting process to include discussing the consent form, verbal consent and thumb-printing.
* Subject has not completed his or her final vaccination in VAC-010.

For Toddlers NOT Enrolled in VAC-010 (PCV-primed-only cohort):

* Healthy Kenyan toddlers between 12 to 15 (inclusive) months of age who have completed their primary Expanded Programme on Immunization (EPI) vaccines, with the exception that the birth dose of oral polio vaccine is not required.
* Subjects who have not received a PCV booster following primary PCV series.
* Subject's parent must provide voluntary written informed consent for subject to participate in the study, is fully capable of comprehending and complying with study requirements and procedures, able and willing to return for all scheduled follow-up visits, and has expressed availability for the required study period, with access to a consistent means of telephone contact. An illiterate parent will require an impartial witness to be present during consenting process to include discussing the consent form, verbal consent and thumb-printing.
* Subjects who were not born premature, had a birth weight of > 2.5 kg, and who have a weight-to-height Z-score of ≥ -2 at the time of enrollment.

Exclusion Criteria:

- For Toddlers NOT enrolled in VAC-010 (PCV-primed only):

* Use of any investigational or non-registered drug within 90 days prior to screening, or planned during the course of study participation.
* Immunosuppression or immunodeficiency (inclusive of human immunodeficiency virus [HIV]) by medical history (inclusive of possible HIV through maternal fetal transfer at time of birth or through breast milk).
* Chronic, clinically significant pulmonary, cardiovascular, hepatobiliary, gastrointestinal, renal, neurological, or hematological functional abnormality or major congenital defects or illness that requires medical therapy, by medical history or clinical assessment. This includes abnormal vital signs as assessed by toxicity scoring.
* Any medical or social condition that in the opinion of the investigator may interfere with the study objectives, pose a risk to the study subject, or prevent the subject from completing the study.
* An employee (or first degree relative of employee) of the Sponsor, the Clinical Research Organization (CRO), the investigator or any site personnel.
* Disorders that required chronic administration (defined as more than 14 consecutive days) of immunosuppressants or other immune-modifying drugs within the 6 months prior to enrollment. An immunosuppressant dose of glucocorticoid will be defined as a systemic dose >10 mg of prednisone (adult dosage) adjusted for equivalent dosing in toddlers by weight. The use of topical glucocorticoids will be permitted.
* Administration of immunoglobulins and/or any blood products within the 6 months preceding enrollment in the study; or anticipation of such administration during the study period.
* History of meningitis, seizures or any neurological disorder.
* Subject who has evidence of congenital abnormality or developmental delay.
* Any evidence of fetal alcohol syndrome or history of alcohol abuse in mother during pregnancy.

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy PCV- primed Kenyan toddlers; some of whom have participated in VAC-010 (n=250) and some of whom have not (n=50)
Sampling Method: Probability Sample
Enrollment: 297 (Actual)
Dates: Start 2014-09-25 (Actual); Primary Completion 2016-02-18 (Actual); Study Completion 2016-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nekoye Otsyula, MB ChB MSc, Principal Investigator — Kenya Medical Research Institute/Walter Reed Project
Locations (1):
- Kenya Medical Research Institute/Walter Reed Project, Kisumu, Kenya

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled healthy Kenyan toddlers who participated in the randomized control trial VAC-010 (NCT02097472) whose parents provided consent to participate in VAC-011. In addition, 50 healthy toddlers who did not participate in the VAC-010 study were enrolled from the community as a pneumococcal conjugate vaccine (PCV)-primed-only open cohort.
Pre-assignment Details: Participants were enrolled sequentially into Cohort 1 (PATH-wSP 300 µg or control) and Cohort 2 (PATH-wSP 600 µg or control).
Period: Overall Study
Arm/Group | PATH-wSP 300 µg + Booster | PATH-wSP 300 µg Only | PATH-wSP 600 µg + Booster | PATH-wSP 600 µg Only | Booster Only (300 µg) | Booster Only (600 µg) | No Intervention (300 µg) | No Intervention (600 µg)
Started | 49 | 49 | 50 | 50 | 24 | 25 | 25 | 25
Completed | 45 | 45 | 43 | 41 | 22 | 24 | 25 | 24
Not Completed | 4 | 4 | 7 | 9 | 2 | 1 | 0 | 1
Not completed — Lost to Follow-up | 2 | 1 | 3 | 3 | 1 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 5 | 1 | 0 | 0 | 0
Not completed — Unable to Comply with Protocol | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Booster Only (Both Cohorts): Toddlers who enrolled in Cohort 1 or Cohort 2 of Study VAC-010 and received one saline injection and the two booster vaccines (Synflorix and Pentavac) followed by a 2nd saline injection 8 weeks later.
- No Intervention: Toddlers who enrolled during Cohort 1 or Cohort 2 who did not participate in Study VAC-010 and did not receive either PATH-wSP or either of the booster vaccines (Pentavac or Synflorix).
- Total: Total of all reporting groups
Arm/Group | PATH-wSP 300 µg + Booster | PATH-wSP 300 µg Only | PATH-wSP 600 µg + Booster | PATH-wSP 600 µg Only | Booster Only (Both Cohorts) | No Intervention | Total
Number analyzed (Participants) | 49 | 49 | 50 | 50 | 49 | 50 | 297
Age, Continuous [Mean (Standard Deviation); unit: months] | 13.2 (1.1) | 13.0 (1.1) | 13.3 (1.1) | 13.5 (1.2) | 13.1 (1.0) | 13.3 (1.2) | 13.2 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 25 | 23 | 24 | 23 | 31 | 157
  Male | 18 | 24 | 27 | 26 | 26 | 19 | 140
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Luhya | 3 | 1 | 7 | 5 | 2 | 1 | 19
  Luo | 45 | 47 | 43 | 45 | 46 | 48 | 274
  Other | 1 | 1 | 0 | 0 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Streptococcus Pneumoniae in Nasopharynx
Description: The prevalence of Streptococcus pneumoniae (SPn) in the nasopharynx was measured by the number (and percentage) of participants positive for SPn detected by quantitative polymerase chain reaction (qPCR) from nasopharyngeal swabs taken at each study visit.
  NPC endpoints were analyzed within combined study groups:
  * PATH-wSP 300 µg: Combines groups who received 300 µg PATH-wSP with or without booster
  * Control (300 µg): Participants in VAC-010 Cohort 1 who received booster-only plus non-interventional participants enrolled during Cohort 1
  * PATH-wSP 600 µg: Combines groups who received 600 µg PATH-wSP with or without booster
  * Control (600 µg): Participants in VAC-010 Cohort 2 who received booster-only plus non-interventional participants enrolled during Cohort 2
Time Frame: Week 0, Week 12, Week 16, Week 20, Week 32
Population: The Nasopharyngeal Carriage (NPC) population included enrolled participants with at least one post-enrollment swab measurement not associated with a protocol violation that may have interfered with the assessment of NPC outcomes. VAC-010 participants who did not receive both vaccinations were excluded.
Measure: Count of Participants; unit: Participants
Groups:
- Combined PATH-wSP 300 µg: All participants who received PATH-wSP 300 µg, including participants in the PATH-wSP 300 µg + Booster and participants in the PATH-wSP 300 µg Only treatment groups.
- Combined Control (300 µg): Participants enrolled during Cohort 1 who received booster-only or no intervention.
- Combined PATH-wSP 600 µg: All participants who received PATH-wSP 600 µg, including participants in the PATH-wSP 600 µg + Booster and participants in the PATH-wSP 600 µg Only treatment groups.
- Combined Control (600 µg): All participants enrolled during Cohort 2 who received booster-only or no intervention.
Arm/Group | Combined PATH-wSP 300 µg | Combined Control (300 µg) | Combined PATH-wSP 600 µg | Combined Control (600 µg)
Number analyzed (Participants) | 91 | 47 | 94 | 50
Participants
  Visit 1 (Week 0): number analyzed (Participants) | 90 | 47 | 94 | 50
  Visit 1 (Week 0) | 76 | 43 | 86 | 46
  Visit 2 (Week 12): number analyzed (Participants) | 90 | 47 | 94 | 50
  Visit 2 (Week 12) | 77 | 44 | 80 | 47
  Visit 3 (Week 16): number analyzed (Participants) | 91 | 47 | 91 | 48
  Visit 3 (Week 16) | 85 | 43 | 81 | 45
  Visit 4 (Week 20): number analyzed (Participants) | 90 | 47 | 88 | 48
  Visit 4 (Week 20) | 85 | 43 | 81 | 44
  Visit 5 (Week 32): number analyzed (Participants) | 89 | 46 | 83 | 48
  Visit 5 (Week 32) | 81 | 43 | 71 | 43

2. Primary Outcome: Density of Streptococcus Pneumoniae in the Nasopharynx
Description: The density of Streptococcus pneumoniae (SPn) in the nasopharynx was measured by the number of autolysin (LytA) gene copies detected by quantitative polymerase chain reaction (qPCR) from nasopharyngeal swabs taken at each study visit.
  NPC endpoints were analyzed within combined study groups:
  * PATH-wSP 300 µg: Combines groups who received 300 µg PATH-wSP with or without booster
  * Control (300 µg): Participants in VAC-010 Cohort 1 who received booster-only plus non-interventional group enrolled during Cohort 1
  * PATH-wSP 600 µg: Combines groups who received 600 µg PATH-wSP with or without booster
  * Control (600 µg): Participants in VAC-010 Cohort 2 who received booster-only, plus non-interventional group enrolled during Cohort 2
Time Frame: Week 0, Week 12, Week 16, Week 20, Week 32
Population: The Nasopharyngeal Carriage (NPC) population with available LytA data at each time point
Measure: Median (95% Confidence Interval); unit: log LytA copies
Arm/Group | Combined PATH-wSP 300 µg | Combined Control (300 µg) | Combined PATH-wSP 600 µg | Combined Control (600 µg)
Number analyzed (Participants) | 79 | 43 | 85 | 49
log LytA copies
  Visit 1 (Week 0): number analyzed (Participants) | 79 | 43 | 81 | 45
  Visit 1 (Week 0) | 13.5 [12.4 to 14.6] | 12.5 [11.7 to 14.4] | 13.9 [13.2 to 14.5] | 13.8 [12.9 to 14.7]
  Visit 2 (Week 12): number analyzed (Participants) | 78 | 39 | 85 | 49
  Visit 2 (Week 12) | 14.0 [12.9 to 14.9] | 13.0 [11.3 to 14.3] | 16.4 [15.6 to 17.2] | 15.9 [14.7 to 17.4]
  Visit 3 (Week 16): number analyzed (Participants) | 78 | 40 | 80 | 40
  Visit 3 (Week 16) | 14.7 [14.0 to 15.2] | 14.5 [13.6 to 15.7] | 16.8 [16.0 to 17.3] | 16.5 [15.2 to 17.5]
  Visit 4 (Week 20): number analyzed (Participants) | 72 | 41 | 81 | 41
  Visit 4 (Week 20) | 15.1 [14.4 to 15.8] | 14.0 [13.1 to 15.2] | 15.5 [14.6 to 16.3] | 15.1 [14.1 to 16.2]
  Visit 5 (Week 32): number analyzed (Participants) | 76 | 39 | 65 | 40
  Visit 5 (Week 32) | 16.8 [16.2 to 17.3] | 14.9 [14.5 to 16.0] | 14.9 [14.1 to 15.7] | 14.8 [14.0 to 15.9]

3. Secondary Outcome: Geometric Mean Concentration (GMC) of Immunoglobulin G (IgG) Antibodies Against Pneumococcal Proteins
Description: Immunogenicity was evaluated based on the following assays:
  1. Immunoglobulin (IgG) response to pneumolysoid [L460D] and pneumococcal surface protein A family 1 [PspA-Fam1] was measured by enzyme-linked immunosorbent assay (ELISA).
  2. IgG response to the following pneumococcal proteins was measured using the Meso Scale Discovery (MSD) platform:
     * L460D
     * PspA-Fam1
     * Pneumococcal histidine triad D (PhtD)
     * Boston Children's Hospital protein 785 (BCH0785)
     * Serine threonine kinase protein (StkP)
     * Pneumococcal choline-binding protein A (PcpA)
     * Streptococcus pneumonia whole cell antigen (SPWCA)
     * Pneumococcal iron uptake protein A (PiuA)
     * Pneumococcal iron acquisition protein A (PiaA)
Time Frame: Baseline (Week 0), 4 weeks post-vaccination 2 (Week 12), and 6 months post-vaccination 2 (Week 32).
Population: The Immunogenicity (IG) population includes participants enrolled in Study VAC-010 with at least one usable value in the VAC-011 immunogenicity data set. VAC-010 participants who did not receive both vaccinations were excluded.
Measure: Geometric Mean (90% Confidence Interval); unit: titer
Arm/Group | PATH-wSP 300 µg + Booster | PATH-wSP 300 µg Only | PATH-wSP 600 µg + Booster | PATH-wSP 600 µg Only | Booster Only (Both Cohorts)
Number analyzed (Participants) | 43 | 40 | 38 | 35 | 38
titer
  Pneumolysoid (L460D): Baseline | 381.12 [272.73 to 532.58] | 330.58 [218.99 to 499.03] | 785.54 [546.78 to 1128.56] | 832.32 [561.77 to 1233.19] | 497.88 [329.88 to 751.44]
  Pneumolysoid (L460D): 4 weeks post-Vaccination 2 | 813.00 [560.96 to 1178.29] | 786.26 [539.05 to 1146.83] | 1600 [1130.57 to 2264.35] | 2330.97 [1571 to 3457.66] | 545.42 [377.42 to 788.21]
  Pneumolysoid (L460D): 6 months post-Vaccination 2 | 1069.31 [739.69 to 1545.80] | 1212.57 [894.84 to 1643.12] | 1372.33 [1021.16 to 1844.25] | 1697.94 [1224.11 to 2355.18] | 1051.76 [757.13 to 1461.05]
  PspA-Fam1 (ELISA): Baseline | 397.94 [284.00 to 557.59] | 382.99 [277.26 to 529.05] | 602.57 [450.01 to 806.85] | 725.31 [533.27 to 986.52] | 513.79 [388.35 to 679.75]
  PspA-Fam1 (ELISA): 4 weeks post-Vaccination 2 | 720.33 [551.98 to 940.03] | 571.29 [418.14 to 780.55] | 870.53 [672.36 to 1127.10] | 1409.82 [979.31 to 2029.60] | 514.81 [362.75 to 730.63]
  PspA-Fam1 (ELISA): 6 months post-Vaccination 2 | 873.74 [618.19 to 1234.94] | 824.96 [558.84 to 1217.81] | 762.72 [555.97 to 1046.35] | 1239.01 [892.62 to 1719.83] | 796.22 [557.37 to 1137.42]
  L460D: Baseline | 261.25 [199.66 to 341.84] | 234.51 [171.83 to 320.05] | 314.86 [240.39 to 412.41] | 346.26 [273.01 to 439.16] | 241.08 [187.27 to 310.35]
  L460D: 4 weeks post-Vaccination 2 | 460.91 [344.59 to 616.50] | 440.19 [335.66 to 577.28] | 622.67 [484.23 to 800.70] | 917.86 [696.84 to 1208.97] | 303.90 [234.88 to 393.22]
  L460D: 6 months post-Vaccination 2 | 499.10 [373.82 to 666.36] | 525.38 [413.09 to 668.18] | 508.30 [384.86 to 671.33] | 701.06 [551.11 to 891.80] | 380.59 [294.18 to 492.39]
  PspA-Fam1 (MSD): Baseline | 172.25 [116.10 to 255.57] | 195.25 [128.65 to 296.33] | 219.55 [151.45 to 318.27] | 231.28 [156.45 to 341.90] | 218.24 [153.16 to 310.99]
  PspA-Fam1 (MSD): 4 weeks post-Vaccination 2 | 368.08 [261.00 to 519.08] | 357.83 [242.60 to 527.79] | 349.00 [254.08 to 479.38] | 609.24 [406.57 to 912.93] | 213.82 [137.75 to 331.91]
  PspA-Fam1 (MSD): 6 months post-Vaccination 2 | 303.31 [208.18 to 441.91] | 339.07 [220.62 to 521.10] | 362.35 [264.93 to 495.58] | 548.93 [383.92 to 784.84] | 317.09 [213.51 to 470.92]
  PhtD: Baseline | 464.43 [335.55 to 642.80] | 456.19 [339.35 to 613.26] | 464.52 [315.74 to 683.42] | 555.72 [415.87 to 742.60] | 377.18 [272.45 to 522.17]
  PhtD: 4 weeks post-Vaccination 2 | 847.28 [636.32 to 1128.18] | 773.24 [610.73 to 979.01] | 702.42 [512.66 to 962.40] | 1174.38 [910.85 to 1514.14] | 575.56 [423.05 to 783.05]
  PhtD: 6 months post-Vaccination 2 | 1128.66 [851.33 to 1496.33] | 1163.21 [946.47 to 1429.57] | 926.31 [692.19 to 1239.60] | 1282.89 [975.69 to 1686.81] | 890.03 [659.09 to 1201.88]
  BCH0785: Baseline | 401.04 [289.77 to 555.05] | 322.75 [239.06 to 435.74] | 267.80 [187.61 to 382.28] | 371.19 [258.34 to 533.31] | 314.85 [213.23 to 464.88]
  BCH0785: 4 weeks post-Vaccination 2 | 555.25 [396.67 to 777.24] | 514.90 [400.37 to 662.18] | 411.22 [297.25 to 568.88] | 761.38 [541.86 to 1069.83] | 397.66 [280.80 to 563.15]
  BCH0785: 6 months post-Vaccination 2 | 539.24 [406.71 to 714.95] | 602.44 [472.33 to 768.40] | 385.46 [279.12 to 532.30] | 726.43 [542.87 to 972.06] | 460.80 [327.57 to 648.21]
  StkP: Baseline | 193.50 [135.62 to 276.08] | 142.90 [107.04 to 190.79] | 163.30 [110.56 to 241.20] | 246.51 [170.96 to 355.45] | 191.77 [136.54 to 269.35]
  StkP: 4 weeks post-Vaccination 2 | 334.14 [238.90 to 467.33] | 240.51 [190.85 to 303.10] | 253.15 [181.99 to 352.13] | 444.83 [322.88 to 612.84] | 235.29 [169.75 to 326.15]
  StkP: 6 months post-Vaccination 2 | 304.48 [219.27 to 422.80] | 331.73 [262.02 to 420.00] | 278.27 [197.74 to 391.60] | 470.92 [345.08 to 642.66] | 305.51 [214.28 to 435.58]
  PcpA: Baseline | 320.15 [199.08 to 514.86] | 369.58 [213.36 to 640.18] | 307.97 [160.95 to 589.28] | 464.90 [278.23 to 776.80] | 302.03 [177.98 to 512.53]
  PcpA: 4 weeks post-Vaccination 2 | 383.75 [237.14 to 620.99] | 358.39 [218.41 to 588.08] | 387.80 [216.85 to 693.50] | 527.74 [303.33 to 918.20] | 351.00 [194.02 to 635.00]
  PcpA: 6 months post-Vaccination 2 | 631.99 [394.03 to 1013.67] | 681.06 [470.01 to 986.87] | 633.57 [400.16 to 1003.12] | 779.77 [499.74 to 1216.72] | 558.79 [338.90 to 921.36]
  SPWCA: Baseline | 676.76 [584.10 to 784.10] | 665.77 [575.42 to 770.30] | 630.23 [527.12 to 753.50] | 669.91 [590.27 to 760.29] | 660.13 [575.51 to 757.18]
  SPWCA: 4 weeks post-Vaccination 2 | 852.45 [735.87 to 987.50] | 782.09 [701.14 to 872.38] | 815.92 [722.01 to 922.06] | 965.60 [817.61 to 1140.38] | 762.31 [663.45 to 875.89]
  SPWCA: 6 months post-Vaccination 2 | 849.99 [730.32 to 989.27] | 908.71 [797.98 to 1034.80] | 828.46 [718.93 to 954.67] | 1020.25 [895.70 to 1162.12] | 700.71 [595.24 to 824.86]
  PiuA: Baseline | 685.69 [530.35 to 886.53] | 631.45 [489.14 to 815.17] | 585.28 [451.15 to 759.30] | 697.84 [521.35 to 934.08] | 608.91 [457.96 to 809.60]
  PiuA: 4 weeks post-Vaccination 2 | 938.09 [717.50 to 1226.49] | 867.54 [693.68 to 1084.98] | 925.23 [758.38 to 1128.79] | 1164.80 [894.83 to 1516.20] | 743.11 [574.02 to 962.00]
  PiuA: 6 months post-Vaccination 2 | 1035.89 [806.39 to 1330.70] | 1274.26 [989.51 to 1640.94] | 998.07 [795.24 to 1252.64] | 1188.92 [927.29 to 1524.37] | 923.97 [665.80 to 1282.27]
  PiaA: Baseline | 650.37 [494.57 to 855.26] | 560.35 [406.33 to 772.74] | 604.16 [453.70 to 804.50] | 886.79 [678.57 to 1158.92] | 606.15 [472.84 to 777.05]
  PiaA: 4 weeks post-Vaccination 2 | 930.90 [705.04 to 1229.10] | 851.40 [651.29 to 1113.01] | 788.37 [626.08 to 992.72] | 1574.97 [1207.40 to 2054.43] | 805.26 [605.90 to 1070.23]
  PiaA: 6 months post-Vaccination | 1014.92 [782.79 to 1315.88] | 1055.71 [782.89 to 1423.60] | 732.05 [556.80 to 962.48] | 1428.92 [1120.44 to 1822.33] | 816.56 [605.56 to 1101.08]

4. Secondary Outcome: Geometric Mean Concentration Ratios of Immunoglobulin G (IgG) Antibodies Against Pneumococcal Proteins for PATH-wSP Groups Versus the Booster Only Group
Description: Data reported are the geometric mean concentration at 6 months post-vaccination 2 (Week 32) for each PATH-wSP group divided by the Booster (Synflorix and Pentavax)-only group (N=38). Immunogenicity was evaluated based on the following assays:
  1. Immunoglobulin (IgG) response to pneumolysoid (L460D) and pneumococcal surface protein A family 1 (PspA-Fam1) was measured by enzyme-linked immunosorbent assay (ELISA).
  2. IgG response to the following pneumococcal proteins was measured using the Meso Scale Discovery (MSD) platform:
     * L460D
     * PspA-Fam1
     * Pneumococcal histidine triad D (PhtD)
     * Boston Children's Hospital protein 785 (BCH0785)
     * Serine threonine kinase protein (StkP)
     * Pneumococcal choline-binding protein A (PcpA)
     * Streptococcus pneumonia whole cell antigen (SPWCA)
     * Pneumococcal iron uptake protein A (PiuA)
     * Pneumococcal iron acquisition protein A (PiaA)
Time Frame: Week 32
Population: Immunogenicity population
Measure: Number (90% Confidence Interval); unit: ratio
Arm/Group | PATH-wSP 300 µg + Booster | PATH-wSP 300 µg Only | PATH-wSP 600 µg + Booster | PATH-wSP 600 µg Only
Number analyzed (Participants) | 43 | 40 | 38 | 35
ratio
  Pneumolysoid (L460D) | 1.02 [0.62 to 1.67] | 1.15 [0.74 to 1.79] | 1.30 [0.84 to 2.02] | 1.61 [1.02 to 2.55]
  PspA-Fam1 (ELISA) | 1.10 [0.67 to 1.79] | 1.04 [0.61 to 1.75] | 0.96 [0.60 to 1.53] | 1.56 [0.96 to 2.52]
  L460D | 1.31 [0.89 to 1.93] | 1.38 [0.98 to 1.95] | 1.34 [0.92 to 1.94] | 1.84 [1.30 to 2.61]
  PspA-Fam1 (MSD) | 0.96 [0.56 to 1.64] | 1.07 [0.60 to 1.91] | 1.14 [0.69 to 1.88] | 1.73 [1.02 to 2.94]
  PhtD | 1.27 [0.84 to 1.91] | 1.31 [0.91 to 1.87] | 1.04 [0.69 to 1.88] | 1.44 [0.96 to 2.16]
  BCH0785 | 1.17 [0.76 to 1.81] | 1.31 [0.87 to 1.97] | 0.84 [0.53 to 1.33] | 1.58 [1.01 to 2.46]
  StkP | 1.00 [0.62 to 1.61] | 1.09 [0.72 to 1.65] | 0.91 [0.56 to 1.48] | 1.54 [0.96 to 2.46]
  PcpA | 1.13 [0.57 to 2.23] | 1.22 [0.66 to 2.24] | 1.13 [0.58 to 2.22] | 1.40 [0.72 to 2.71]
  SPWCA | 1.21 [0.97 to 1.51] | 1.30 [1.06 to 1.59] | 1.18 [0.96 to 1.46] | 1.46 [1.18 to 1.79]
  PiuA | 1.12 [0.75 to 1.68] | 1.38 [0.92 to 2.07] | 1.08 [0.73 to 1.60] | 1.29 [0.85 to 1.94]
  PiaA | 1.24 [0.84 to 1.83] | 1.29 [0.85 to 1.96] | 0.90 [0.60 to 1.34] | 1.75 [1.19 to 2.57]

5. Secondary Outcome: Geometric Mean Fold Change of Immunoglobulin G (IgG) Antibodies Against Pneumococcal Proteins
Description: Immunogenicity was evaluated based on the following assays:
  1. IgG response to pneumolysoid [L460D] and pneumococcal surface protein A family 1 [PspA-Fam1] was measured by enzyme-linked immunosorbent assay (ELISA).
  2. IgG response to the following pneumococcal proteins was measured using the Meso Scale Discovery (MSD) platform:
     * L460D
     * PspA-Fam1
     * Pneumococcal histidine triad D (PhtD)
     * Boston Children's Hospital protein 785 (BCH0785)
     * Serine threonine kinase protein (StkP)
     * Pneumococcal choline-binding protein A (PcpA)
     * Streptococcus pneumonia whole cell antigen (SPWCA)
     * Pneumococcal iron uptake protein A (PiuA)
     * Pneumococcal iron acquisition protein A (PiaA)
  The fold-change was calculated as the 6-month post-vaccination (Week 32) IgG response divided by the Baseline IgG response.
Time Frame: Baseline and Week 32
Population: Immunogenicity Population
Measure: Geometric Mean (90% Confidence Interval); unit: fold-change
Arm/Group | PATH-wSP 300 µg + Booster | PATH-wSP 300 µg Only | PATH-wSP 600 µg + Booster | PATH-wSP 600 µg Only | Booster Only (Both Cohorts)
Number analyzed (Participants) | 43 | 40 | 38 | 35 | 38
fold-change
  Pneumolysoid (L460D) | 2.81 [2.09 to 3.76] | 3.67 [2.88 to 4.67] | 1.75 [1.36 to 2.24] | 2.04 [1.54 to 2.69] | 2.11 [1.47 to 3.03]
  PspA-Fam1 (ELISA) | 2.20 [1.64 to 2.94] | 2.15 [1.50 to 3.10] | 1.27 [0.89 to 1.81] | 1.71 [1.20 to 2.43] | 1.55 [1.15 to 2.08]
  L460D | 1.91 [1.51 to 2.42] | 2.24 [1.81 to 2.78] | 1.61 [1.27 to 2.04] | 2.02 [1.64 to 2.50] | 1.58 [1.25 to 1.99]
  PspA-Fam1 (MSD) | 1.76 [1.25 to 2.49] | 1.74 [1.13 to 2.66] | 1.65 [1.17 to 2.32] | 2.37 [1.64 to 3.44] | 1.45 [1.05 to 2.02]
  PhtD | 2.43 [1.87 to 3.16] | 2.55 [1.96 to 3.31] | 1.99 [1.48 to 2.68] | 2.31 [1.81 to 2.95] | 2.36 [1.77 to 3.15]
  BCH0785 | 1.34 [1.04 to 1.73] | 1.87 [1.48 to 2.36] | 1.44 [1.10 to 1.88] | 1.96 [1.49 to 2.46] | 1.59 [1.28 to 1.98]
  StkP | 1.57 [1.17 to 2.11] | 2.32 [1.80 to 2.99] | 1.70 [1.32 to 2.19] | 1.91 [1.48 to 2.46] | 1.59 [1.28 to 1.98]
  PcpA | 1.97 [1.44 to 2.71] | 1.84 [1.16 to 2.94] | 2.06 [1.36 to 3.12] | 1.68 [1.19 to 2.36] | 1.85 [1.19 to 2.88]
  SPWCA | 1.26 [1.04 to 1.52] | 1.36 [1.17 to 1.59] | 1.31 [1.11 to 1.56] | 1.52 [1.35 to 1.72] | 1.06 [0.88 to 1.28]
  PiuA | 1.51 [1.22 to 1.88] | 2.02 [1.62 to 2.51] | 1.71 [1.32 to 2.20] | 1.70 [1.38 to 2.10] | 1.52 [1.24 to 1.85]
  PiaA | 1.56 [1.18 to 2.07] | 1.88 [1.39 to 2.56] | 1.21 [0.99 to 1.49] | 1.61 [1.23 to 2.12] | 1.35 [1.03 to 1.76]

6. Secondary Outcome: Percentage of Participants Meeting Seroresponse Fold-Rise Categories at 6 Months Post Vaccination 2
Description: The percentage of participants with a seroresponse, defined as a ≥ 2, ≥ 3, and ≥ 4 fold-rise above Baseline in IgG antibody levels against Pneumococcal proteins. Fold-rise was calculated as the 6-month post-vaccination (Week 32) IgG response divided by the Baseline IgG level.
  Immunogenicity was evaluated based on the following assays:
  1. IgG response to pneumolysoid [L460D] and pneumococcal surface protein A family 1 [PspA-Fam1] was measured by enzyme-linked immunosorbent assay (ELISA).
  2. IgG response to the following pneumococcal proteins was measured using the Meso Scale Discovery (MSD) platform:
     * L460D
     * PspA-Fam1
     * Pneumococcal histidine triad D (PhtD)
     * Boston Children's Hospital protein 785 (BCH0785)
     * Serine threonine kinase protein (StkP)
     * Pneumococcal choline-binding protein A (PcpA)
     * Streptococcus pneumonia whole cell antigen (SPWCA)
     * Pneumococcal iron uptake protein A (PiuA)
     * Pneumococcal iron acquisition protein A (PiaA)
Time Frame: Baseline and Week 32
Population: Immunogenicity Population
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | PATH-wSP 300 µg + Booster | PATH-wSP 300 µg Only | PATH-wSP 600 µg + Booster | PATH-wSP 600 µg Only | Booster Only (Both Cohorts)
Number analyzed (Participants) | 43 | 40 | 38 | 35 | 38
percentage of participants
  Pneumolysoid (L460D): ≥ 2 Fold-Rise | 72.1 [58.74 to 83.04] | 87.5 [75.50 to 94.94] | 60.5 [45.90 to 73.86] | 62.9 [47.56 to 76.44] | 55.3 [40.75 to 69.13]
  Pneumolysoid (L460D): ≥ 3 Fold-Rise | 44.2 [31.20 to 57.80] | 57.5 [43.31 to 70.82] | 28.9 [17.16 to 43.33] | 34.3 [21.12 to 49.55] | 39.5 [26.14 to 54.10]
  Pneumolysoid (L460D): ≥4 Fold-Rise | 44.2 [31.20 to 57.80] | 57.5 [43.31 to 70.82] | 26.3 [15.03 to 40.54] | 34.3 [21.12 to 49.55] | 39.5 [26.14 to 54.10]
  PspA-Fam1 (ELISA): ≥ 2 Fold-Rise | 41.9 [29.08 to 55.52] | 60.0 [45.78 to 73.06] | 28.9 [17.16 to 43.33] | 42.9 [28.58 to 58.08] | 36.8 [23.83 to 51.47]
  PspA-Fam1 (ELISA): ≥ 3 Fold-Rise | 32.6 [20.88 to 46.13] | 42.5 [29.18 to 56.69] | 15.8 [7.11 to 28.80] | 37.1 [23.56 to 52.44] | 26.3 [15.03 to 40.54]
  PspA-Fam1 (ELISA): ≥ 4 Fold-Rise | 25.6 [15.06 to 38.77] | 30.0 [18.31 to 44.03] | 13.2 [5.33 to 25.70] | 22.9 [11.91 to 37.48] | 23.7 [12.95 to 37.69]
  L460D: ≥ 2 Fold-Rise | 46.5 [33.35 to 60.05] | 52.5 [38.48 to 66.23] | 34.2 [21.56 to 48.80] | 48.6 [33.79 to 63.54] | 36.8 [23.83 to 51.47]
  L460D: ≥ 3 Fold-Rise | 23.3 [13.20 to 36.25] | 40.0 [26.94 to 54.22] | 15.8 [7.11 to 28.80] | 31.4 [18.73 to 46.61] | 18.4 [8.98 to 31.83]
  L460D: ≥ 4 Fold-Rise | 14.0 [6.26 to 25.69] | 27.5 [16.25 to 41.39] | 10.5 [3.68 to 22.49] | 17.1 [7.74 to 31.06] | 10.5 [3.68 to 22.49]
  PspA-Fam1 (MSD): ≥ 2 Fold-Rise | 32.6 [20.88 to 46.13] | 37.5 [24.73 to 51.72] | 44.7 [30.87 to 59.25] | 45.7 [31.17 to 60.83] | 39.5 [26.14 to 54.10]
  PspA-Fam1 (MSD): ≥ 3 Fold-Rise | 25.6 [15.06 to 38.77] | 30.0 [18.31 to 44.03] | 31.6 [19.34 to 46.09] | 42.9 [28.58 to 58.08] | 21.1 [10.93 to 34.79]
  PspA-Fam1 (MSD): ≥ 4 Fold-Rise | 20.9 [11.38 to 33.68] | 27.5 [16.25 to 41.39] | 23.7 [12.95 to 37.69] | 31.4 [18.73 to 46.61] | 15.8 [7.11 to 28.80]
  PhtD: ≥ 2 Fold-Ris2 | 58.1 [44.48 to 70.92] | 50.0 [36.11 to 63.89] | 57.9 [43.31 to 71.52] | 54.3 [39.17 to 68.83] | 60.5 [45.90 to 73.86]
  PhtD: ≥ 3 Fold-Rise | 46.5 [33.35 to 60.05] | 40.0 [26.94 to 54.22] | 28.9 [17.16 to 43.33] | 40.0 [26.05 to 55.28] | 42.1 [28.48 to 56.69]
  PhtD: ≥ 4 Fold-Rise | 25.6 [15.06 to 37.77] | 35.0 [22.55 to 49.49] | 15.8 [7.11 to 28.80] | 17.1 [7.74 to 31.06] | 28.9 [17.16 to 43.33]
  BCH0785: ≥ 2 Fold-Rise | 32.6 [20.88 to 46.13] | 50.0 [36.11 to 63.89] | 42.1 [28.48 to 56.69] | 42.9 [28.58 to 58.08] | 39.5 [26.14 to 54.10]
  BCH0785: ≥ 3 Fold-Rise | 23.3 [13.20 to 36.25] | 27.5 [16.25 to 41.39] | 18.4 [8.98 to 31.83] | 28.6 [16.40 to 43.63] | 26.3 [15.03 to 40.54]
  BCH0785: ≥ 4 Fold-Rise | 14.0 [6.26 to 25.69] | 15.0 [6.74 to 27.47] | 10.5 [3.68 to 22.49] | 25.7 [14.12 to 40.58] | 15.8 [7.11 to 28.80]
  StkP: ≥ 2 Fold-Rise | 32.6 [20.88 to 46.13] | 52.5 [38.48 to 66.23] | 42.1 [28.48 to 56.69] | 48.06 [33.79 to 63.54] | 36.8 [23.83 to 51.47]
  StkP: ≥ 3 Fold-Rise | 20.9 [11.38 to 33.68] | 32.5 [20.41 to 46.63] | 23.7 [12.95 to 37.69] | 34.3 [21.12 to 49.55] | 21.1 [10.93 to 34.79]
  StkP: ≥ 4 Fold-Rise | 18.6 [9.61 to 31.07] | 27.5 [16.25 to 41.39] | 10.5 [3.68 to 22.49] | 20.0 [9.78 to 34.30] | 13.2 [5.33 to 25.70]
  PcpA: ≥ 2 Fold-Rise | 46.5 [33.35 to 60.05] | 42.5 [29.18 to 56.69] | 50.0 [35.74 to 64.26] | 40.0 [26.05 to 55.28] | 39.5 [26.14 to 54.10]
  PcpA: ≥ 3 Fold-Rise | 30.2 [18.90 to 43.71] | 35.0 [22.55 to 49.19] | 34.2 [21.56 to 48.80] | 31.4 [18.73 to 46.61] | 31.6 [19.34 to 46.09]
  PcpA: ≥ 4 Fold-Rise | 25.6 [15.06 to 38.77] | 27.5 [16.25 to 41.39] | 26.3 [15.03 to 40.54] | 22.9 [11.91 to 37.48] | 31.6 [19.34 to 46.09]
  SPWCA: ≥ 2 Fold-Rise | 25.6 [15.06 to 38.77] | 22.5 [12.27 to 35.98] | 26.3 [15.03 to 40.54] | 31.4 [18.73 to 46.61] | 21.1 [10.93 to 34.79]
  SPWCA: ≥ 3 Fold-Rise | 9.3 [3.24 to 20.04] | 12.5 [5.06 to 24.50] | 10.5 [3.68 to 22.49] | 2.9 [0.15 to 12.85] | 2.6 [0.13 to 11.89]
  SPWCA: ≥ 4 Fold-Rise | 4.7 [0.83 to 13.93] | 7.5 [2.08 to 18.26] | 0.0 [0.00 to 7.58] | 0.0 [0.00 to 8.20] | 2.6 [0.13 to 11.89]
  PiuA: ≥ 2 Fold-Rise | 32.6 [20.88 to 46.13] | 52.5 [38.48 to 66.23] | 39.5 [26.14 to 54.10] | 45.7 [31.17 to 60.83] | 34.2 [21.56 to 48.80]
  PiuA: ≥ 3 Fold-Rise | 20.9 [11.38 to 33.68] | 27.5 [16.25 to 41.39] | 26.3 [15.03 to 40.54] | 22.9 [11.91 to 37.48] | 13.2 [5.33 to 25.70]
  PiuA: ≥ 4 Fold-Rise | 9.3 [3.24 to 20.04] | 22.5 [12.27 to 35.98] | 15.8 [7.11 to 28.80] | 17.1 [7.74 to 31.06] | 7.9 [2.19 to 19.16]
  PiaA: ≥ 2 Fold-Rise | 41.9 [29.08 to 55.52] | 40.0 [26.94 to 54.22] | 26.3 [15.03 to 40.54] | 40.0 [26.05 to 55.28] | 36.8 [23.83 to 51.47]
  PiaA: ≥ 3 Fold-Rise | 23.3 [13.20 to 36.25] | 25.0 [14.24 to 38.71] | 7.9 [2.19 to 19.16] | 20.0 [9.78 to 34.30] | 21.1 [10.93 to 34.79]
  PiaA: ≥ 4 Fold-Rise | 11.6 [4.70 to 22.91] | 20.0 [10.36 to 33.20] | 2.6 [0.13 to 11.89] | 17.1 [7.74 to 31.06] | 10.5 [3.68 to 22.49]

7. Secondary Outcome: Number of Participants With Neutralizing Antibody Response to Pneumolysin
Description: Neutralizing antibody responses to pneumolysin were assessed at Baseline and 6 months post vaccination 2 using an in vitro toxin neutralization assay that measures the ability of antibodies to neutralize wild-type pneumolysin-induced lysis of rabbit red blood cells.
  Each sample was categorized as negative (< 1/20 dilution) or positive (with titer between 1/20 and 1/320 dilution). Responses at higher dilutions indicate higher levels of neutralizing antibodies to pneumolysin.
Time Frame: Baseline (Week 0) and 6 months post-vaccination 2 (Week 32)
Population: Immunogenicity Population with available neutralizing antibody data.
Measure: Count of Participants; unit: Participants
Arm/Group | PATH-wSP 300 µg + Booster | PATH-wSP 300 µg Only | PATH-wSP 600 µg + Booster | PATH-wSP 600 µg Only | Booster Only (Both Cohorts)
Number analyzed (Participants) | 35 | 34 | 37 | 35 | 34
Participants
  Baseline: <1:20 titer | 12 | 10 | 12 | 8 | 17
  Baseline: 1:20 titer | 10 | 10 | 11 | 8 | 8
  Baseline: 1:40 titer | 8 | 8 | 9 | 12 | 4
  Baseline: 1:80 titer | 2 | 5 | 3 | 6 | 4
  Baseline: 1:160 titer | 1 | 0 | 2 | 1 | 1
  Baseline: 1:320 titer | 2 | 1 | 0 | 0 | 0
  6 months post-vaccination 2: <1:20 titer | 0 | 0 | 0 | 0 | 0
  6 months post-vaccination 2: 1:20 titer | 11 | 12 | 11 | 7 | 12
  6 months post-vaccination 2: 1:40 titer | 10 | 11 | 12 | 8 | 12
  6 months post-vaccination 2: 1:80 titer | 5 | 5 | 8 | 10 | 7
  6 months post-vaccination 2: 1:160 titer | 7 | 5 | 4 | 7 | 3
  6 months post-vaccination 2: 1:320 titer | 2 | 1 | 2 | 3 | 0

8. Secondary Outcome: Number of Adverse Events (AE)
Description: An AE was defined as any untoward, undesired, or unplanned event in the form of signs, symptoms, disease, or laboratory or psychological/physiologic observations occurring in a person in a clinical study. The AEs collected in this non-interventional study were those that remained open after the last visit in the VAC-010 Study, those attributed to study vaccine in VAC-010 with onset after the participant exited VAC-010, those that were related to a VAC-011 procedure (i.e. blood draw, nasal swab sample), and all serious adverse events.
Time Frame: 32 weeks; for participants enrolled concurrently in Study VAC-010 adverse events were collected after the last VAC-010 visit through to Week 32.
Population: All enrolled participants
Measure: Number; unit: adverse events
Arm/Group | PATH-wSP 300 µg + Booster | PATH-wSP 300 µg Only | PATH-wSP 600 µg + Booster | PATH-wSP 600 µg Only | Booster Only (Both Cohorts) | No Intervention
Number analyzed (Participants) | 49 | 49 | 50 | 50 | 49 | 50
adverse events
  Total number of AEs | 0 | 0 | 1 | 4 | 1 | 1
  Serious AE: No | 0 | 0 | 1 | 0 | 0 | 0
  Serious AE: Yes | 0 | 0 | 0 | 4 | 1 | 1
  Severity: Mild (Grade 1) | 0 | 0 | 1 | 0 | 0 | 1
  Severity: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0
  Severity: Severe (Grade 3) | 0 | 0 | 0 | 4 | 1 | 1
  Severity: Potentially Life Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Severity: Death (Grade 5) | 0 | 0 | 0 | 0 | 0 | 0
  Related to vaccine: No | 0 | 0 | 1 | 4 | 1 | 1
  Related to vaccine: Yes | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Prevalence of Streptococcus Pneumoniae Serotype 11A/D/E [11A] in the Nasopharynx
Description: Nasopharyngeal samples were further analyzed for the prevalence of specific Streptococcus pneumoniae serotypes by microarray. The number of participants with a positive result for SPn serotype 11A/D/E [11A] is reported.
  NPC endpoints were analyzed within combined study groups:
  * PATH-wSP 300 µg: Combines groups who received 300 µg PATH-wSP with or without booster
  * Control (300 µg): Participants in VAC-010 Cohort 1 who received booster-only, plus non-interventional group enrolled during Cohort 1
  * PATH-wSP 600 µg: Combines groups who received 600 µg PATH-wSP with or without booster
  * Control (600 µg): Participants in VAC-010 Cohort 2 who received booster-only, plus non-interventional group enrolled during Cohort 2
Time Frame: Week 0, Week 12, Week 16, Week 20, Week 32
Population: Nasopharyngeal Carriage (NPC) population with culture-confirmed samples and available serotype data at each time point
Measure: Count of Participants; unit: Participants
Arm/Group | Combined PATH-wSP 300 µg | Combined Control (300 µg) | Combined PATH-wSP 600 µg | Combined Control (600 µg)
Number analyzed (Participants) | 81 | 43 | 83 | 50
Participants
  Visit 1 (Week 0): number analyzed (Participants) | 81 | 43 | 83 | 42
  Visit 1 (Week 0) | 6 | 4 | 6 | 1
  Visit 2 (Week 12): number analyzed (Participants) | 79 | 40 | 83 | 50
  Visit 2 (Week 12) | 7 | 3 | 5 | 1
  Visit 3 (Week 16): number analyzed (Participants) | 77 | 38 | 80 | 40
  Visit 3 (Week 16) | 2 | 4 | 7 | 3
  Visit 4 (Week 20): number analyzed (Participants) | 73 | 41 | 81 | 42
  Visit 4 (Week 20) | 4 | 3 | 5 | 1
  Visit 5 (Week 32): number analyzed (Participants) | 74 | 39 | 63 | 39
  Visit 5 (Week 32) | 6 | 0 | 9 | 3

10. Secondary Outcome: Prevalence of Streptococcus Pneumoniae Serotype 13 in the Nasopharynx
Description: Nasopharyngeal samples were further analyzed for the prevalence of specific Streptococcus pneumoniae serotypes by microarray. The number of participants with a positive result for SPn serotype 13 is reported.
  NPC endpoints were analyzed within combined study groups:
  * PATH-wSP 300 µg: Combines groups who received 300 µg PATH-wSP with or without booster
  * Control (300 µg): Participants in VAC-010 Cohort 1 who received booster-only, plus non-interventional group enrolled during Cohort 1
  * PATH-wSP 600 µg: Combines groups who received 600 µg PATH-wSP with or without booster
  * Control (600 µg): Participants in VAC-010 Cohort 2 who received booster-only, plus non-interventional group enrolled during Cohort 2
Time Frame: Week 0, Week 12, Week 16, Week 20, Week 32
Population: Nasopharyngeal Carriage (NPC) population with culture-confirmed samples and available serotype data at each time point
Measure: Count of Participants; unit: Participants
Arm/Group | Combined PATH-wSP 300 µg | Combined Control (300 µg) | Combined PATH-wSP 600 µg | Combined Control (600 µg)
Number analyzed (Participants) | 83 | 43 | 85 | 50
Participants
  Visit 1 (Week 0): number analyzed (Participants) | 81 | 43 | 83 | 42
  Visit 1 (Week 0) | 6 | 2 | 3 | 5
  Visit 2 (Week 12): number analyzed (Participants) | 79 | 40 | 83 | 49
  Visit 2 (Week 12) | 6 | 5 | 5 | 3
  Visit 3 (Week 16): number analyzed (Participants) | 78 | 38 | 81 | 40
  Visit 3 (Week 16) | 4 | 3 | 5 | 1
  Visit 4 (Week 20): number analyzed (Participants) | 73 | 41 | 81 | 42
  Visit 4 (Week 20) | 6 | 5 | 5 | 1
  Visit 5 (Week 32): number analyzed (Participants) | 74 | 39 | 63 | 39
  Visit 5 (Week 32) | 5 | 6 | 4 | 2

11. Secondary Outcome: Prevalence of Streptococcus Pneumoniae Serotype 15A in the Nasopharynx
Description: Nasopharyngeal samples were further analyzed for the prevalence of specific Streptococcus pneumoniae serotypes by microarray. The number of participants with a positive result for SPn serotype 15A is reported.
  NPC endpoints were analyzed within combined study groups:
  * PATH-wSP 300 µg: Combines groups who received 300 µg PATH-wSP with or without booster
  * Control (300 µg): Participants in VAC-010 Cohort 1 who received booster-only, plus non-interventional group enrolled during Cohort 1
  * PATH-wSP 600 µg: Combines groups who received 600 µg PATH-wSP with or without booster
  * Control (600 µg): Participants in VAC-010 Cohort 2 who received booster-only, plus non-interventional group enrolled during Cohort 2
Time Frame: Week 0, Week 12, Week 16, Week 20, Week 32
Population: Nasopharyngeal Carriage (NPC) population with culture-confirmed samples and available serotype data at each time point
Measure: Count of Participants; unit: Participants
Arm/Group | Combined PATH-wSP 300 µg | Combined Control (300 µg) | Combined PATH-wSP 600 µg | Combined Control (600 µg)
Number analyzed (Participants) | 83 | 43 | 85 | 50
Participants
  Visit 1 (Week 0): number analyzed (Participants) | 83 | 43 | 83 | 42
  Visit 1 (Week 0) | 1 | 0 | 2 | 3
  Visit 2 (Week 12): number analyzed (Participants) | 79 | 40 | 83 | 49
  Visit 2 (Week 12) | 5 | 2 | 5 | 4
  Visit 3 (Week 16): number analyzed (Participants) | 78 | 38 | 81 | 40
  Visit 3 (Week 16) | 8 | 1 | 5 | 1
  Visit 4 (Week 20): number analyzed (Participants) | 73 | 42 | 81 | 42
  Visit 4 (Week 20) | 7 | 1 | 6 | 2
  Visit 5 (Week 32): number analyzed (Participants) | 74 | 39 | 63 | 39
  Visit 5 (Week 32) | 7 | 4 | 2 | 5

12. Secondary Outcome: Prevalence of Streptococcus Pneumoniae Serotype 15B/C [15B] in the Nasopharynx
Description: Nasopharyngeal samples were further analyzed for the prevalence of specific Streptococcus pneumoniae serotypes by microarray. The number of participants with a positive result for SPn serotype 15B/C [15B] is reported.
  NPC endpoints were analyzed within combined study groups:
  * PATH-wSP 300 µg: Combines groups who received 300 µg PATH-wSP with or without booster
  * Control (300 µg): Participants in VAC-010 Cohort 1 who received booster-only, plus non-interventional group enrolled during Cohort 1
  * PATH-wSP 600 µg: Combines groups who received 600 µg PATH-wSP with or without booster
  * Control (600 µg): Participants in VAC-010 Cohort 2 who received booster-only, plus non-interventional group enrolled during Cohort 2
Time Frame: Week 0, Week 12, Week 16, Week 20, Week 32
Population: Nasopharyngeal Carriage (NPC) population with culture-confirmed samples and available serotype data at each time point
Measure: Count of Participants; unit: Participants
Arm/Group | Combined PATH-wSP 300 µg | Combined Control (300 µg) | Combined PATH-wSP 600 µg | Combined Control (600 µg)
Number analyzed (Participants) | 83 | 43 | 85 | 50
Participants
  Visit 1 (Week 0): number analyzed (Participants) | 81 | 43 | 83 | 42
  Visit 1 (Week 0) | 10 | 2 | 9 | 6
  Visit 2 (Week 12): number analyzed (Participants) | 79 | 40 | 84 | 49
  Visit 2 (Week 12) | 16 | 3 | 7 | 5
  Visit 3 (Week 16): number analyzed (Participants) | 78 | 38 | 81 | 40
  Visit 3 (Week 16) | 9 | 4 | 5 | 8
  Visit 4 (Week 20): number analyzed (Participants) | 73 | 41 | 81 | 42
  Visit 4 (Week 20) | 11 | 2 | 9 | 4
  Visit 5 (Week 32): number analyzed (Participants) | 74 | 38 | 63 | 39
  Visit 5 (Week 32) | 4 | 1 | 4 | 3

13. Secondary Outcome: Prevalence of Streptococcus Pneumoniae Serotype 19A in the Nasopharynx
Description: Nasopharyngeal samples were further analyzed for the prevalence of specific Streptococcus pneumoniae serotypes by microarray. The number of participants with a positive result for SPn serotype 19A is reported.
  NPC endpoints were analyzed within combined study groups:
  * PATH-wSP 300 µg: Combines groups who received 300 µg PATH-wSP with or without booster
  * Control (300 µg): Participants in VAC-010 Cohort 1 who received booster-only, plus non-interventional group enrolled during Cohort 1
  * PATH-wSP 600 µg: Combines groups who received 600 µg PATH-wSP with or without booster
  * Control (600 µg): Participants in VAC-010 Cohort 2 who received booster-only, plus non-interventional group enrolled during Cohort 2
Time Frame: Week 0, Week 12, Week 16, Week 20, Week 32
Population: Nasopharyngeal Carriage (NPC) population with culture-confirmed samples and available serotype data at each time point
Measure: Count of Participants; unit: Participants
Arm/Group | Combined PATH-wSP 300 µg | Combined Control (300 µg) | Combined PATH-wSP 600 µg | Combined Control (600 µg)
Number analyzed (Participants) | 83 | 43 | 85 | 50
Participants
  Visit 1 (Week 0): number analyzed (Participants) | 81 | 43 | 83 | 42
  Visit 1 (Week 0) | 3 | 4 | 7 | 4
  Visit 2 (Week 12): number analyzed (Participants) | 79 | 40 | 84 | 49
  Visit 2 (Week 12) | 3 | 6 | 9 | 5
  Visit 3 (Week 16): number analyzed (Participants) | 77 | 38 | 80 | 40
  Visit 3 (Week 16) | 1 | 7 | 6 | 3
  Visit 4 (Week 20): number analyzed (Participants) | 74 | 41 | 81 | 42
  Visit 4 (Week 20) | 2 | 6 | 5 | 6
  Visit 5 (Week 32): number analyzed (Participants) | 74 | 39 | 63 | 39
  Visit 5 (Week 32) | 7 | 3 | 3 | 4

14. Secondary Outcome: Prevalence of Streptococcus Pneumoniae Serotype 19F in the Nasopharynx
Description: Nasopharyngeal samples were further analyzed for the prevalence of specific Streptococcus pneumoniae serotypes by microarray. The number of participants with a positive result for SPn serotype 19F is reported.
  NPC endpoints were analyzed within combined study groups:
  * PATH-wSP 300 µg: Combines groups who received 300 µg PATH-wSP with or without booster
  * Control (300 µg): Participants in VAC-010 Cohort 1 who received booster-only, plus non-interventional group enrolled during Cohort 1
  * PATH-wSP 600 µg: Combines groups who received 600 µg PATH-wSP with or without booster
  * Control (600 µg): Participants in VAC-010 Cohort 2 who received booster-only, plus non-interventional group enrolled during Cohort 2
Time Frame: Week 0, Week 12, Week 16, Week 20, Week 32
Population: Nasopharyngeal Carriage (NPC) population with culture-confirmed samples and available serotype data at each time point
Measure: Count of Participants; unit: Participants
Arm/Group | Combined PATH-wSP 300 µg | Combined Control (300 µg) | Combined PATH-wSP 600 µg | Combined Control (600 µg)
Number analyzed (Participants) | 83 | 43 | 85 | 50
Participants
  Visit 1 (Week 0): number analyzed (Participants) | 82 | 43 | 83 | 42
  Visit 1 (Week 0) | 4 | 2 | 6 | 5
  Visit 2 (Week 12): number analyzed (Participants) | 79 | 40 | 84 | 49
  Visit 2 (Week 12) | 5 | 5 | 7 | 3
  Visit 3 (Week 16): number analyzed (Participants) | 78 | 38 | 80 | 40
  Visit 3 (Week 16) | 4 | 5 | 10 | 2
  Visit 4 (Week 20): number analyzed (Participants) | 74 | 41 | 81 | 42
  Visit 4 (Week 20) | 5 | 4 | 10 | 3
  Visit 5 (Week 32): number analyzed (Participants) | 74 | 39 | 63 | 39
  Visit 5 (Week 32) | 4 | 3 | 8 | 2

15. Secondary Outcome: Prevalence of Streptococcus Pneumoniae Serotype 3 in the Nasopharynx
Description: Nasopharyngeal samples were further analyzed for the prevalence of specific Streptococcus pneumoniae serotypes by microarray. The number of participants with a positive result for SPn serotype 3 is reported.
  NPC endpoints were analyzed within combined study groups:
  * PATH-wSP 300 µg: Combines groups who received 300 µg PATH-wSP with or without booster
  * Control (300 µg): Participants in VAC-010 Cohort 1 who received booster-only, plus non-interventional group enrolled during Cohort 1
  * PATH-wSP 600 µg: Combines groups who received 600 µg PATH-wSP with or without booster
  * Control (600 µg): Participants in VAC-010 Cohort 2 who received booster-only, plus non-interventional group enrolled during Cohort 2
Time Frame: Week 0, Week 12, Week 16, Week 20, Week 32
Population: Nasopharyngeal Carriage (NPC) population with culture-confirmed samples and available serotype data at each time point
Measure: Count of Participants; unit: Participants
Arm/Group | Combined PATH-wSP 300 µg | Combined Control (300 µg) | Combined PATH-wSP 600 µg | Combined Control (600 µg)
Number analyzed (Participants) | 83 | 43 | 85 | 50
Participants
  Visit 1 (Week 0): number analyzed (Participants) | 81 | 43 | 83 | 42
  Visit 1 (Week 0) | 8 | 4 | 5 | 2
  Visit 2 (Week 12): number analyzed (Participants) | 79 | 40 | 84 | 50
  Visit 2 (Week 12) | 6 | 4 | 7 | 1
  Visit 3 (Week 16): number analyzed (Participants) | 78 | 38 | 80 | 40
  Visit 3 (Week 16) | 9 | 4 | 11 | 2
  Visit 4 (Week 20): number analyzed (Participants) | 73 | 41 | 81 | 42
  Visit 4 (Week 20) | 6 | 5 | 6 | 4
  Visit 5 (Week 32): number analyzed (Participants) | 74 | 39 | 63 | 38
  Visit 5 (Week 32) | 4 | 4 | 8 | 1

16. Secondary Outcome: Prevalence of Streptococcus Pneumoniae Serotype 35B in the Nasopharynx
Description: Nasopharyngeal samples were further analyzed for the prevalence of specific Streptococcus pneumoniae serotypes by microarray. The number of participants with a positive result for SPn serotype 35B is reported.
  NPC endpoints were analyzed within combined study groups:
  * PATH-wSP 300 µg: Combines groups who received 300 µg PATH-wSP with or without booster
  * Control (300 µg): Participants in VAC-010 Cohort 1 who received booster-only, plus non-interventional group enrolled during Cohort 1
  * PATH-wSP 600 µg: Combines groups who received 600 µg PATH-wSP with or without booster
  * Control (600 µg): Participants in VAC-010 Cohort 2 who received booster-only, plus non-interventional group enrolled during Cohort 2
Time Frame: Week 0, Week 12, Week 16, Week 20, Week 32
Population: Nasopharyngeal Carriage (NPC) population with culture-confirmed samples and available serotype data at each time point
Measure: Count of Participants; unit: Participants
Arm/Group | Combined PATH-wSP 300 µg | Combined Control (300 µg) | Combined PATH-wSP 600 µg | Combined Control (600 µg)
Number analyzed (Participants) | 83 | 43 | 85 | 50
Participants
  Visit 1 (Week 0): number analyzed (Participants) | 81 | 43 | 83 | 42
  Visit 1 (Week 0) | 8 | 4 | 11 | 4
  Visit 2 (Week 12): number analyzed (Participants) | 79 | 40 | 84 | 49
  Visit 2 (Week 12) | 8 | 3 | 9 | 4
  Visit 3 (Week 16): number analyzed (Participants) | 78 | 38 | 80 | 40
  Visit 3 (Week 16) | 5 | 6 | 8 | 2
  Visit 4 (Week 20): number analyzed (Participants) | 74 | 41 | 81 | 42
  Visit 4 (Week 20) | 2 | 5 | 6 | 3
  Visit 5 (Week 32): number analyzed (Participants) | 74 | 39 | 63 | 38
  Visit 5 (Week 32) | 7 | 3 | 4 | 1

17. Secondary Outcome: Prevalence of Streptococcus Pneumoniae Serotype 6A/B [6A] in the Nasopharynx
Description: Nasopharyngeal samples were further analyzed for the prevalence of specific Streptococcus pneumoniae serotypes by microarray. The number of participants with a positive result for SPn serotype 6A/B [6A] is reported.
  NPC endpoints were analyzed within combined study groups:
  * PATH-wSP 300 µg: Combines groups who received 300 µg PATH-wSP with or without booster
  * Control (300 µg): Participants in VAC-010 Cohort 1 who received booster-only, plus non-interventional group enrolled during Cohort 1
  * PATH-wSP 600 µg: Combines groups who received 600 µg PATH-wSP with or without booster
  * Control (600 µg): Participants in VAC-010 Cohort 2 who received booster-only, plus non-interventional group enrolled during Cohort 2
Time Frame: Week 0, Week 12, Week 16, Week 20, Week 32
Population: Nasopharyngeal Carriage (NPC) population with culture-confirmed samples and available serotype data at each time point
Measure: Count of Participants; unit: Participants
Arm/Group | Combined PATH-wSP 300 µg | Combined Control (300 µg) | Combined PATH-wSP 600 µg | Combined Control (600 µg)
Number analyzed (Participants) | 83 | 43 | 85 | 50
Participants
  Visit 1 (Week 0): number analyzed (Participants) | 81 | 43 | 83 | 42
  Visit 1 (Week 0) | 5 | 5 | 6 | 2
  Visit 2 (Week 12): number analyzed (Participants) | 79 | 40 | 85 | 49
  Visit 2 (Week 12) | 7 | 4 | 6 | 3
  Visit 3 (Week 16): number analyzed (Participants) | 78 | 38 | 80 | 40
  Visit 3 (Week 16) | 5 | 6 | 7 | 1
  Visit 4 (Week 20): number analyzed (Participants) | 73 | 41 | 81 | 42
  Visit 4 (Week 20) | 3 | 3 | 5 | 3
  Visit 5 (Week 32): number analyzed (Participants) | 74 | 39 | 63 | 39
  Visit 5 (Week 32) | 4 | 5 | 5 | 2

18. Secondary Outcome: Prevalence of Streptococcus Pneumoniae Serotype NT4b in the Nasopharynx
Description: Nasopharyngeal samples were further analyzed for the prevalence of specific Streptococcus pneumoniae serotypes by microarray. The number of participants with a positive result for SPn serotype NT4b is reported.
  NPC endpoints were analyzed within combined study groups:
  * PATH-wSP 300 µg: Combines groups who received 300 µg PATH-wSP with or without booster
  * Control (300 µg): Participants in VAC-010 Cohort 1 who received booster-only, plus non-interventional group enrolled during Cohort 1
  * PATH-wSP 600 µg: Combines groups who received 600 µg PATH-wSP with or without booster
  * Control (600 µg): Participants in VAC-010 Cohort 2 who received booster-only, plus non-interventional group enrolled during Cohort 2
Time Frame: Week 0, Week 12, Week 16, Week 20, Week 32
Population: Nasopharyngeal Carriage (NPC) population with culture-confirmed samples and available serotype data at each time point
Measure: Count of Participants; unit: Participants
Arm/Group | Combined PATH-wSP 300 µg | Combined Control (300 µg) | Combined PATH-wSP 600 µg | Combined Control (600 µg)
Number analyzed (Participants) | 83 | 43 | 85 | 50
Participants
  Visit 1 (Week 0): number analyzed (Participants) | 81 | 43 | 83 | 42
  Visit 1 (Week 0) | 29 | 17 | 27 | 15
  Visit 2 (Week 12): number analyzed (Participants) | 79 | 40 | 84 | 49
  Visit 2 (Week 12) | 17 | 10 | 32 | 10
  Visit 3 (Week 16): number analyzed (Participants) | 78 | 38 | 80 | 40
  Visit 3 (Week 16) | 17 | 13 | 23 | 10
  Visit 4 (Week 20): number analyzed (Participants) | 73 | 41 | 81 | 42
  Visit 4 (Week 20) | 12 | 15 | 26 | 8
  Visit 5 (Week 32): number analyzed (Participants) | 74 | 39 | 63 | 39
  Visit 5 (Week 32) | 20 | 14 | 18 | 13

19. Secondary Outcome: Density of Streptococcus Pneumoniae Serotype 11A/D/E [11A] in the Nasopharynx
Description: The density of Streptococcus pneumoniae serotype 11A/D/E [11A] in the nasopharynx was measured by the number of LytA gene copies detected by microarray from nasopharyngeal swabs taken at each study visit.
  NPC endpoints were analyzed within combined study groups:
  * PATH-wSP 300 µg: Combines groups who received 300 µg PATH-wSP with or without booster
  * Control (300 µg): Participants in VAC-010 Cohort 1 who received booster-only, plus non-interventional group enrolled during Cohort 1
  * PATH-wSP 600 µg: Combines groups who received 600 µg PATH-wSP with or without booster
  * Control (600 µg): Participants in VAC-010 Cohort 2 who received booster-only, plus non-interventional group enrolled during Cohort 2
Time Frame: Week 0, Week 12, Week 16, Week 20, Week 32
Population: NPC population with culture-confirmed samples and a relative abundance greater than zero for the serotype.
Measure: Median (95% Confidence Interval); unit: log LytA copies
Arm/Group | Combined PATH-wSP 300 µg | Combined Control (300 µg) | Combined PATH-wSP 600 µg | Combined Control (600 µg)
Number analyzed (Participants) | 7 | 4 | 9 | 3
log LytA copies
  Visit 1 (Week 0): number analyzed (Participants) | 6 | 4 | 6 | 1
  Visit 1 (Week 0) | 11.9 [10.2 to 13.6] | 15.0 [9.8 to 16.7] | 12.9 [3.2 to 16.7] | 14 [14.0 to 14.0]
  Visit 2 (Week 12): number analyzed (Participants) | 7 | 3 | 5 | 1
  Visit 2 (Week 12) | 10.9 [7.1 to 15.3] | 17.6 [11.9 to 19.7] | 14.4 [12.3 to 15.7] | 18.5 [18.5 to 18.5]
  Visit 3 (Week 16): number analyzed (Participants) | 2 | 4 | 7 | 3
  Visit 3 (Week 16) | 9.8 [9.4 to 10.3] | 13.6 [11.5 to 14.9] | 16.6 [14.7 to 21.3] | 14.1 [9.0 to 16.9]
  Visit 4 (Week 20): number analyzed (Participants) | 4 | 3 | 5 | 1
  Visit 4 (Week 20) | 15.1 [13.9 to 22.3] | 12.3 [10.5 to 13.4] | 15.8 [13.3 to 20.3] | 5.4 [5.4 to 5.4]
  Visit 5 (Week 32): number analyzed (Participants) | 6 | 0 | 9 | 3
  Visit 5 (Week 32) | 16.3 [16.1 to 19.9] |  | 14.5 [11.1 to 17.3] | 16.4 [14.5 to 17.1]

20. Secondary Outcome: Density of Streptococcus Pneumoniae Serotype 13 in the Nasopharynx
Description: The density of Streptococcus pneumoniae serotype 13 in the nasopharynx was measured by the number of LytA gene copies detected by microarray from nasopharyngeal swabs taken at each study visit.
  NPC endpoints were analyzed within combined study groups:
  * PATH-wSP 300 µg: Combines groups who received 300 µg PATH-wSP with or without booster
  * Control (300 µg): Participants in VAC-010 Cohort 1 who received booster-only, plus non-interventional group enrolled during Cohort 1
  * PATH-wSP 600 µg: Combines groups who received 600 µg PATH-wSP with or without booster
  * Control (600 µg): Participants in VAC-010 Cohort 2 who received booster-only, plus non-interventional group enrolled during Cohort 2
Time Frame: Week 0, Week 12, Week 16, Week 20, Week 32
Population: NPC population with culture-confirmed samples and a relative abundance greater than zero for the serotype.
Measure: Median (95% Confidence Interval); unit: log LytA copies
Arm/Group | Combined PATH-wSP 300 µg | Combined Control (300 µg) | Combined PATH-wSP 600 µg | Combined Control (600 µg)
Number analyzed (Participants) | 6 | 6 | 5 | 5
log LytA copies
  Visit 1 (Week 0): number analyzed (Participants) | 6 | 2 | 3 | 5
  Visit 1 (Week 0) | 12.9 [9.8 to 15.0] | 17.1 [7.0 to 17.1] | 12.2 [9.8 to 13.8] | 12.3 [10.0 to 18.6]
  Visit 2 (Week 12): number analyzed (Participants) | 6 | 5 | 5 | 3
  Visit 2 (Week 12) | 10.6 [5.1 to 16.1] | 11.6 [5.7 to 14.3] | 15.0 [3.0 to 17.3] | 12.1 [10.3 to 15.8]
  Visit 3 (Week 16): number analyzed (Participants) | 4 | 3 | 5 | 1
  Visit 3 (Week 16) | 14.2 [10.7 to 17.7] | 15.6 [12.9 to 19.3] | 17.7 [14.0 to 20.3] | 13.8 [13.8 to 13.8]
  Visit 4 (Week 20): number analyzed (Participants) | 6 | 5 | 5 | 1
  Visit 4 (Week 20) | 13.2 [10.7 to 16.7] | 13.1 [11.6 to 14.0] | 13.4 [11.6 to 18.7] | 14.6 [14.6 to 14.6]
  Visit 5 (Week 32): number analyzed (Participants) | 5 | 6 | 4 | 2
  Visit 5 (Week 32) | 14.5 [11.4 to 19.0] | 14.7 [10.2 to 15.1] | 15.8 [10.0 to 22.3] | 16.2 [13.8 to 18.5]

21. Secondary Outcome: Density of Streptococcus Pneumoniae Serotype 15A in the Nasopharynx
Description: The density of Streptococcus pneumoniae serotype 15A in the nasopharynx was measured by the number of LytA gene copies detected by microarray from nasopharyngeal swabs taken at each study visit.
  NPC endpoints were analyzed within combined study groups:
  * PATH-wSP 300 µg: Combines groups who received 300 µg PATH-wSP with or without booster
  * Control (300 µg): Participants in VAC-010 Cohort 1 who received booster-only, plus non-interventional group enrolled during Cohort 1
  * PATH-wSP 600 µg: Combines groups who received 600 µg PATH-wSP with or without booster
  * Control (600 µg): Participants in VAC-010 Cohort 2 who received booster-only, plus non-interventional group enrolled during Cohort 2
Time Frame: Week 0, Week 12, Week 16, Week 20, Week 32
Population: NPC population with culture-confirmed samples and a relative abundance greater than zero for the serotype.
Measure: Median (95% Confidence Interval); unit: log LytA copies
Arm/Group | Combined PATH-wSP 300 µg | Combined Control (300 µg) | Combined PATH-wSP 600 µg | Combined Control (600 µg)
Number analyzed (Participants) | 8 | 4 | 6 | 5
log LytA copies
  Visit 1 (Week 0): number analyzed (Participants) | 1 | 0 | 2 | 3
  Visit 1 (Week 0) | 13.7 [13.7 to 13.7] |  | 16.1 [15.1 to 17.2] | 11.0 [9.8 to 13.4]
  Visit 2 (Week 12): number analyzed (Participants) | 5 | 2 | 5 | 4
  Visit 2 (Week 12) | 14.1 [11.3 to 16.0] | 13.8 [11.2 to 16.3] | 18.5 [15.6 to 18.7] | 16.3 [11.7 to 19.2]
  Visit 3 (Week 16): number analyzed (Participants) | 8 | 1 | 5 | 1
  Visit 3 (Week 16) | 14.1 [12.4 to 17.2] | 12.3 [12.3 to 12.3] | 15.8 [13.2 to 16.8] | 18.9 [18.9 to 18.9]
  Visit 4 (Week 20): number analyzed (Participants) | 7 | 1 | 6 | 2
  Visit 4 (Week 20) | 13.7 [11.2 to 16.8] | 13.1 [13.1 to 13.1] | 13.7 [11.8 to 16.2] | 15.8 [13.8 to 17.9]
  Visit 5 (Week 32): number analyzed (Participants) | 7 | 4 | 2 | 5
  Visit 5 (Week 32) | 18.0 [14.5 to 19.2] | 16.3 [14.2 to 21.3] | 15.2 [14.8 to 15.6] | 12.9 [9.2 to 19.9]

22. Secondary Outcome: Density of Streptococcus Pneumoniae Serotype 15B/C [15B] in the Nasopharynx
Description: The density of Streptococcus pneumoniae serotype 15B/C [15B] in the nasopharynx was measured by the number of LytA gene copies detected by microarray from nasopharyngeal swabs taken at each study visit.
  NPC endpoints were analyzed within combined study groups:
  * PATH-wSP 300 µg: Combines groups who received 300 µg PATH-wSP with or without booster
  * Control (300 µg): Participants in VAC-010 Cohort 1 who received booster-only, plus non-interventional group enrolled during Cohort 1
  * PATH-wSP 600 µg: Combines groups who received 600 µg PATH-wSP with or without booster
  * Control (600 µg): Participants in VAC-010 Cohort 2 who received booster-only, plus non-interventional group enrolled during Cohort 2
Time Frame: Week 0, Week 12, Week 16, Week 20, Week 32
Population: NPC population with culture-confirmed samples and a relative abundance greater than zero for the serotype.
Measure: Median (95% Confidence Interval); unit: log LytA copies
Arm/Group | Combined PATH-wSP 300 µg | Combined Control (300 µg) | Combined PATH-wSP 600 µg | Combined Control (600 µg)
Number analyzed (Participants) | 16 | 4 | 9 | 8
log LytA copies
  Visit 1 (Week 0): number analyzed (Participants) | 10 | 2 | 9 | 6
  Visit 1 (Week 0) | 13.2 [11.5 to 14.6] | 10.3 [8.7 to 11.9] | 12.1 [9.8 to 15.6] | 14.7 [10.9 to 16.5]
  Visit 2 (Week 12): number analyzed (Participants) | 16 | 3 | 7 | 5
  Visit 2 (Week 12) | 13.0 [10.9 to 15.0] | 10.4 [8.3 to 15.8] | 15.8 [14.7 to 17.2] | 17.9 [16.3 to 19.3]
  Visit 3 (Week 16): number analyzed (Participants) | 9 | 4 | 5 | 8
  Visit 3 (Week 16) | 13.7 [11.4 to 15.7] | 13.5 [12.9 to 16.4] | 20.0 [16.5 to 20.9] | 17.3 [14.4 to 18.9]
  Visit 4 (Week 20): number analyzed (Participants) | 11 | 2 | 9 | 4
  Visit 4 (Week 20) | 13.9 [11.7 to 16.4] | 17.5 [14.9 to 20.2] | 14.9 [11.1 to 17.2] | 17.2 [12.3 to 19.2]
  Visit 5 (Week 32): number analyzed (Participants) | 4 | 1 | 4 | 3
  Visit 5 (Week 32) | 16.7 [14.8 to 20.2] | 17.3 [17.3 to 17.3] | 11.2 [3.7 to 15.7] | 12.8 [10.6 to 13.9]

23. Secondary Outcome: Density of Streptococcus Pneumoniae Serotype 19A in the Nasopharynx
Description: The density of Streptococcus pneumoniae serotype 19A in the nasopharynx was measured by the number of LytA gene copies detected by microarray from nasopharyngeal swabs taken at each study visit.
  NPC endpoints were analyzed within combined study groups:
  * PATH-wSP 300 µg: Combines groups who received 300 µg PATH-wSP with or without booster
  * Control (300 µg): Participants in VAC-010 Cohort 1 who received booster-only, plus non-interventional group enrolled during Cohort 1
  * PATH-wSP 600 µg: Combines groups who received 600 µg PATH-wSP with or without booster
  * Control (600 µg): Participants in VAC-010 Cohort 2 who received booster-only, plus non-interventional group enrolled during Cohort 2
Time Frame: Week 0, Week 12, Week 16, Week 20, Week 32
Population: NPC population with culture-confirmed samples and a relative abundance greater than zero for the serotype.
Measure: Median (95% Confidence Interval); unit: log LytA copies
Arm/Group | Combined PATH-wSP 300 µg | Combined Control (300 µg) | Combined PATH-wSP 600 µg | Combined Control (600 µg)
Number analyzed (Participants) | 7 | 7 | 9 | 6
log LytA copies
  Visit 1 (Week 0): number analyzed (Participants) | 3 | 4 | 7 | 4
  Visit 1 (Week 0) | 10.3 [6.4 to 15.7] | 12.9 [8.7 to 15.2] | 12.3 [11.4 to 14.6] | 11.0 [7.4 to 15.3]
  Visit 2 (Week 12): number analyzed (Participants) | 3 | 6 | 9 | 5
  Visit 2 (Week 12) | 14.2 [5.2 to 15.3] | 12.3 [9.9 to 13.5] | 16.9 [11.3 to 18.6] | 15.5 [11.4 to 19.6]
  Visit 3 (Week 16): number analyzed (Participants) | 1 | 7 | 6 | 3
  Visit 3 (Week 16) | 15.1 [15.1 to 15.1] | 10.6 [7.0 to 16.0] | 16.7 [13.2 to 17.7] | 14.6 [13.6 to 14.9]
  Visit 4 (Week 20): number analyzed (Participants) | 2 | 6 | 5 | 6
  Visit 4 (Week 20) | 18.1 [16.0 to 20.2] | 15.3 [8.7 to 18.2] | 13.3 [12.0 to 17.0] | 14.9 [7.8 to 19.5]
  Visit 5 (Week 32): number analyzed (Participants) | 7 | 3 | 3 | 4
  Visit 5 (Week 32) | 17.0 [13.7 to 19.2] | 15.2 [13.0 to 22.4] | 12.2 [5.4 to 16.8] | 12.9 [5.8 to 20.0]

24. Secondary Outcome: Density of Streptococcus Pneumoniae Serotype 19F in the Nasopharynx
Description: The density of Streptococcus pneumoniae serotype 19F in the nasopharynx was measured by the number of LytA gene copies detected by microarray from nasopharyngeal swabs taken at each study visit.
  NPC endpoints were analyzed within combined study groups:
  * PATH-wSP 300 µg: Combines groups who received 300 µg PATH-wSP with or without booster
  * Control (300 µg): Participants in VAC-010 Cohort 1 who received booster-only, plus non-interventional group enrolled during Cohort 1
  * PATH-wSP 600 µg: Combines groups who received 600 µg PATH-wSP with or without booster
  * Control (600 µg): Participants in VAC-010 Cohort 2 who received booster-only, plus non-interventional group enrolled during Cohort 2
Time Frame: Week 0, Week 12, Week 16, Week 20, Week 32
Population: NPC population with culture-confirmed samples and a relative abundance greater than zero for the serotype.
Measure: Median (95% Confidence Interval); unit: log LytA copies
Arm/Group | Combined PATH-wSP 300 µg | Combined Control (300 µg) | Combined PATH-wSP 600 µg | Combined Control (600 µg)
Number analyzed (Participants) | 5 | 5 | 10 | 5
log LytA copies
  Visit 1 (Week 0): number analyzed (Participants) | 4 | 2 | 6 | 5
  Visit 1 (Week 0) | 14.6 [13.4 to 16.4] | 12.2 [10.6 to 13.8] | 12.7 [11.1 to 16.2] | 12.9 [12.3 to 20.0]
  Visit 2 (Week 12): number analyzed (Participants) | 5 | 5 | 7 | 3
  Visit 2 (Week 12) | 13.3 [12.1 to 17.8] | 13.7 [13.0 to 15.3] | 12.2 [11.6 to 17.5] | 18.2 [10.1 to 19.7]
  Visit 3 (Week 16): number analyzed (Participants) | 4 | 5 | 10 | 2
  Visit 3 (Week 16) | 14.6 [10.2 to 17.7] | 13.0 [11.8 to 17.9] | 16.1 [14.4 to 17.4] | 9.9 [5.8 to 13.9]
  Visit 4 (Week 20): number analyzed (Participants) | 5 | 4 | 10 | 3
  Visit 4 (Week 20) | 12.8 [5.4 to 15.4] | 14.9 [11.5 to 19.7] | 16.7 [13.9 to 17.9] | 11.1 [10.1 to 12.6]
  Visit 5 (Week 32): number analyzed (Participants) | 4 | 3 | 8 | 2
  Visit 5 (Week 32) | 14.6 [10.6 to 17.8] | 17.7 [7.7 to 17.9] | 15.3 [13.7 to 17.1] | 14.1 [13.3 to 14.8]

25. Secondary Outcome: Density of Streptococcus Pneumoniae Serotype 3 in the Nasopharynx
Description: The density of Streptococcus pneumoniae serotype 3 in the nasopharynx was measured by the number of LytA gene copies detected by microarray from nasopharyngeal swabs taken at each study visit.
  NPC endpoints were analyzed within combined study groups:
  * PATH-wSP 300 µg: Combines groups who received 300 µg PATH-wSP with or without booster
  * Control (300 µg): Participants in VAC-010 Cohort 1 who received booster-only, plus non-interventional group enrolled during Cohort 1
  * PATH-wSP 600 µg: Combines groups who received 600 µg PATH-wSP with or without booster
  * Control (600 µg): Participants in VAC-010 Cohort 2 who received booster-only, plus non-interventional group enrolled during Cohort 2
Time Frame: Week 0, Week 12, Week 16, Week 20, Week 32
Population: NPC population with culture-confirmed samples and a relative abundance greater than zero for the serotype.
Measure: Median (95% Confidence Interval); unit: log LytA copies
Arm/Group | Combined PATH-wSP 300 µg | Combined Control (300 µg) | Combined PATH-wSP 600 µg | Combined Control (600 µg)
Number analyzed (Participants) | 9 | 5 | 11 | 4
log LytA copies
  Visit 1 (Week 0): number analyzed (Participants) | 8 | 4 | 5 | 2
  Visit 1 (Week 0) | 12.7 [10.7 to 14.2] | 11.1 [3.7 to 14.7] | 9.7 [8.3 to 15.6] | 12.4 [7.7 to 15.0]
  Visit 2 (Week 12): number analyzed (Participants) | 6 | 4 | 7 | 1
  Visit 2 (Week 12) | 14.2 [10.9 to 18.6] | 11.0 [8.4 to 14.3] | 16.4 [13.5 to 17.9] | 13.3 [13.3 to 13.3]
  Visit 3 (Week 16): number analyzed (Participants) | 9 | 4 | 11 | 2
  Visit 3 (Week 16) | 13.9 [11.2 to 15.7] | 12.7 [11.3 to 15.9] | 15.2 [14.1 to 16.7] | 15.4 [14.8 to 16.1]
  Visit 4 (Week 20): number analyzed (Participants) | 6 | 5 | 6 | 4
  Visit 4 (Week 20) | 13.3 [10.9 to 17.5] | 14.1 [11.8 to 15.5] | 14.7 [13.6 to 19.4] | 17.9 [12.5 to 20.6]
  Visit 5 (Week 32): number analyzed (Participants) | 4 | 4 | 8 | 1
  Visit 5 (Week 32) | 14.6 [12.0 to 19.7] | 14.2 [11.4 to 17.0] | 13.6 [11.0 to 17.4] | 16.6 [16.6 to 16.6]

26. Secondary Outcome: Density of Streptococcus Pneumoniae Serotype 35B in the Nasopharynx
Description: The density of Streptococcus pneumoniae serotype 35B in the nasopharynx was measured by the number of LytA gene copies detected by microarray from nasopharyngeal swabs taken at each study visit.
  NPC endpoints were analyzed within combined study groups:
  * PATH-wSP 300 µg: Combines groups who received 300 µg PATH-wSP with or without booster
  * Control (300 µg): Participants in VAC-010 Cohort 1 who received booster-only, plus non-interventional group enrolled during Cohort 1
  * PATH-wSP 600 µg: Combines groups who received 600 µg PATH-wSP with or without booster
  * Control (600 µg): Participants in VAC-010 Cohort 2 who received booster-only, plus non-interventional group enrolled during Cohort 2
Time Frame: Week 0, Week 12, Week 16, Week 20, Week 32
Population: NPC population with culture-confirmed samples and a relative abundance greater than zero for the serotype.
Measure: Median (95% Confidence Interval); unit: log LytA copies
Arm/Group | Combined PATH-wSP 300 µg | Combined Control (300 µg) | Combined PATH-wSP 600 µg | Combined Control (600 µg)
Number analyzed (Participants) | 8 | 6 | 11 | 4
log LytA copies
  Visit 1 (Week 0): number analyzed (Participants) | 8 | 4 | 11 | 4
  Visit 1 (Week 0) | 14.1 [11.1 to 16.0] | 11.1 [8.5 to 13.0] | 13.1 [10.8 to 14.7] | 12.3 [11.2 to 13.4]
  Visit 2 (Week 12): number analyzed (Participants) | 8 | 3 | 9 | 4
  Visit 2 (Week 12) | 14.3 [9.0 to 15.1] | 9.1 [8.4 to 17.8] | 14.0 [9.7 to 17.2] | 14.3 [11.7 to 16.0]
  Visit 3 (Week 16): number analyzed (Participants) | 5 | 6 | 8 | 2
  Visit 3 (Week 16) | 13.8 [8.3 to 15.5] | 15.5 [13.1 to 18.4] | 15.3 [12.1 to 19.3] | 19.3 [17.9 to 20.8]
  Visit 4 (Week 20): number analyzed (Participants) | 2 | 5 | 6 | 3
  Visit 4 (Week 20) | 8.6 [2.0 to 15.3] | 16.8 [12.4 to 18.5] | 12.8 [11.4 to 15.4] | 11.7 [1.5 to 16.1]
  Visit 5 (Week 32): number analyzed (Participants) | 7 | 3 | 4 | 1
  Visit 5 (Week 32) | 16.0 [10.2 to 18.0] | 13.4 [12.8 to 18.4] | 14.5 [11.3 to 16.4] | 12.2 [12.2 to 12.2]

27. Secondary Outcome: Density of Streptococcus Pneumoniae Serotype 6A/B [6A] in the Nasopharynx
Description: The density of Streptococcus pneumoniae serotype 6A/B [6A] in the nasopharynx was measured by the number of LytA gene copies detected by microarray from nasopharyngeal swabs taken at each study visit.
  NPC endpoints were analyzed within combined study groups:
  * PATH-wSP 300 µg: Combines groups who received 300 µg PATH-wSP with or without booster
  * Control (300 µg): Participants in VAC-010 Cohort 1 who received booster-only, plus non-interventional group enrolled during Cohort 1
  * PATH-wSP 600 µg: Combines groups who received 600 µg PATH-wSP with or without booster
  * Control (600 µg): Participants in VAC-010 Cohort 2 who received booster-only, plus non-interventional group enrolled during Cohort 2
Time Frame: Week 0, Week 12, Week 16, Week 20, Week 32
Population: NPC population with culture-confirmed samples and a relative abundance greater than zero for the serotype.
Measure: Median (95% Confidence Interval); unit: log LytA copies
Arm/Group | Combined PATH-wSP 300 µg | Combined Control (300 µg) | Combined PATH-wSP 600 µg | Combined Control (600 µg)
Number analyzed (Participants) | 7 | 6 | 7 | 3
log LytA copies
  Visit 1 (Week 0): number analyzed (Participants) | 5 | 5 | 6 | 2
  Visit 1 (Week 0) | 14.5 [7.1 to 17.6] | 12.4 [9.0 to 14.5] | 13.4 [11.4 to 14.3] | 11.6 [10.1 to 13.2]
  Visit 2 (Week 12): number analyzed (Participants) | 7 | 4 | 6 | 3
  Visit 2 (Week 12) | 15.0 [13.2 to 18.9] | 12.6 [8.1 to 14.6] | 14.7 [9.6 to 17.2] | 15.8 [1.5 to 16.7]
  Visit 3 (Week 16): number analyzed (Participants) | 5 | 6 | 7 | 1
  Visit 3 (Week 16) | 14.6 [11.9 to 17.5] | 15.0 [10.6 to 18.0] | 14.9 [12.3 to 19.5] | 14.8 [14.8 to 14.8]
  Visit 4 (Week 20): number analyzed (Participants) | 3 | 3 | 5 | 3
  Visit 4 (Week 20) | 20.5 [16.9 to 21.5] | 11.7 [3.1 to 12.6] | 16.6 [9.3 to 17.9] | 12.7 [12.2 to 18.7]
  Visit 5 (Week 32): number analyzed (Participants) | 4 | 5 | 5 | 2
  Visit 5 (Week 32) | 17.2 [14.7 to 17.3] | 14.9 [11.4 to 19.1] | 14.5 [8.3 to 16.4] | 12.6 [11.3 to 14.0]

28. Secondary Outcome: Density of Streptococcus Pneumoniae Serotype NT4b in the Nasopharynx
Description: The density of Streptococcus pneumoniae serotype NT4b in the nasopharynx was measured by the number of LytA gene copies detected by microarray from nasopharyngeal swabs taken at each study visit.
  NPC endpoints were analyzed within combined study groups:
  * PATH-wSP 300 µg: Combines groups who received 300 µg PATH-wSP with or without booster
  * Control (300 µg): Participants in VAC-010 Cohort 1 who received booster-only, plus non-interventional group enrolled during Cohort 1
  * PATH-wSP 600 µg: Combines groups who received 600 µg PATH-wSP with or without booster
  * Control (600 µg): Participants in VAC-010 Cohort 2 who received booster-only, plus non-interventional group enrolled during Cohort 2
Time Frame: Week 0, Week 12, Week 16, Week 20, Week 32
Population: NPC population with culture-confirmed samples and a relative abundance greater than zero for the serotype.
Measure: Median (95% Confidence Interval); unit: log LytA copies
Arm/Group | Combined PATH-wSP 300 µg | Combined Control (300 µg) | Combined PATH-wSP 600 µg | Combined Control (600 µg)
Number analyzed (Participants) | 29 | 17 | 32 | 15
log LytA copies
  Visit 1 (Week 0): number analyzed (Participants) | 29 | 17 | 27 | 15
  Visit 1 (Week 0) | 11.7 [8.5 to 13.7] | 9.8 [8.2 to 12.5] | 10.7 [9.9 to 13.1] | 11.7 [9.4 to 13.1]
  Visit 2 (Week 12): number analyzed (Participants) | 17 | 10 | 32 | 10
  Visit 2 (Week 12) | 12.1 [9.1 to 14.8] | 12.2 [9.8 to 12.9] | 13.4 [12.4 to 14.9] | 12.1 [7.7 to 15.0]
  Visit 3 (Week 16): number analyzed (Participants) | 17 | 13 | 23 | 10
  Visit 3 (Week 16) | 11.7 [9.8 to 13.7] | 12.1 [9.7 to 14.5] | 13.7 [11.2 to 14.5] | 13.7 [11.1 to 15.9]
  Visit 4 (Week 20): number analyzed (Participants) | 12 | 15 | 26 | 8
  Visit 4 (Week 20) | 12.4 [10.0 to 14.3] | 9.6 [8.5 to 12.0] | 12.1 [10.1 to 13.6] | 11.5 [9.7 to 13.1]
  Visit 5 (Week 32): number analyzed (Participants) | 20 | 14 | 18 | 13
  Visit 5 (Week 32) | 14.2 [12.9 to 16.6] | 11.7 [9.8 to 13.2] | 12.1 [9.1 to 13.3] | 12.2 [10.5 to 13.0]

ADVERSE EVENTS:
Time Frame: 32 weeks; for participants enrolled concurrently in Study VAC-010 adverse events were collected after the last VAC-010 visit through to Week 32.
Description: The AEs collected in this non-interventional study were those that remained open after the last visit in the VAC-010 Study, those attributed to study vaccine in VAC-010 with onset after the participant exited VAC-010, those that were related to a VAC-011 procedure (i.e. blood draw, nasal swab sample), and all serious adverse events.
Arm/Group | PATH-wSP 300 µg + Booster | PATH-wSP 300 µg Only | PATH-wSP 600 µg + Booster | PATH-wSP 600 µg Only | Booster Only (Both Cohorts) | No Intervention
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49 | 0/50 | 0/50 | 0/49 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49 | 0/50 | 3/50 | 1/49 | 1/50
Other Adverse Events (participants affected / at risk) | 0/49 | 0/49 | 1/50 | 0/50 | 0/49 | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PATH-wSP 300 µg + Booster (N=49) | PATH-wSP 300 µg Only (N=49) | PATH-wSP 600 µg + Booster (N=50) | PATH-wSP 600 µg Only (N=50) | Booster Only (Both Cohorts) (N=49) | No Intervention (N=50)
Cerebral malaria (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Malaria (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PATH-wSP 300 µg + Booster (N=49) | PATH-wSP 300 µg Only (N=49) | PATH-wSP 600 µg + Booster (N=50) | PATH-wSP 600 µg Only (N=50) | Booster Only (Both Cohorts) (N=49) | No Intervention (N=50)
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No